CLINICAL TRIAL: NCT01775800
Title: Treatment Modification and Symptom Burden in High-Risk Dialysis Patients
Brief Title: Treatment Modification to Reduce Symptom Burden in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1207012494
Record Dates: First submitted 2013-01-16; First posted 2013-01-25 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment modification (Experimental): Patients in this arm will be treated to different targets of blood pressure, parathyroid hormone and serum phosphorus.
  Interventions: Other: Treatment modification
- Usual care (No Intervention): Patients will receive the usual hemodialysis care with no modifications

INTERVENTIONS:
Other: Treatment modification
  Arms: Treatment modification

SUMMARY:
Many patients on hemodialysis experience high rates of symptom burden, such as pain, depression, anxiety and difficulty breathing. This study seeks to reduce these symptoms by modifying the usual guidelines used to manage patients on hemodialysis. For example, rather than trying to keep serum phosphorus below 5.5, patients enrolled in this study may have treatment goals of less than 6.5, in order to reduce the number of pills they need to take and potentially reduce harmful side effects. Blood pressure and serum parathyroid hormone goals will also be modified, to see if these modifications help hemodialysis patients feel better.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patient
* transplant ineligible

Exclusion Criteria:

* dementia
* unable to answer questionnaires for any reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Berman, M.D., Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

REFERENCES:
- [Result] Berman N, Reid MC, Teresi J, Eimicke JP, Adelman R. More with Less: A Trial of Reduced-Intensity Treatment in Transplant-Ineligible Hemodialysis Patients. J Palliat Med. 2016 May;19(5):503-8. doi: 10.1089/jpm.2015.0338. PMID 27139523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 300 dialysis patients screened. 51 were eligible to participate and 16 were randomized.
Groups:
- Treatment Modification: Patients in this arm will be treated to different targets of blood pressure, parathyroid hormone and serum phosphorus.
  Treatment modification
Period: Overall Study
Arm/Group | Treatment Modification | Usual Care
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Modification: Patients were treated to modified goals in terms of blood pressure, parathyroid hormone and phosphorus
- Usual Care: Patients were treated to traditional goals in terms of blood pressure, parathyroid hormone and phosphorus
- Total: Total of all reporting groups
Arm/Group | Treatment Modification | Usual Care | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.38 (10.29) | 69.50 (16.59) | 70.94 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited, Consented, Randomized and Completed
Time Frame: Each participant was assessed for 6 weeks; total recruitment period was 15 months
Population: This number represents the entire dialysis population
Measure: Count of Participants; unit: Participants
Groups:
- Dialysis Patients: Patients were recruited from two dialysis units, one located in Manhattan and on in Queens, New York, representing the total dialysis population
Arm/Group | Dialysis Patients
Number analyzed (Participants) | 300
Participants
  Transplant ineligible | 51
  Consented | 16
  Data collected | 16
  Completed | 16

2. Secondary Outcome: Symptom Burden
Description: Number of symptoms in past week as measured by the Dialysis Symptom Index
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: symptoms
Arm/Group | Treatment Modification | Usual Care
Number analyzed (Participants) | 8 | 8
symptoms
  Baseline | 9.00 (5.45) | 13.25 (6.88)
  6 weeks | 11.00 (6.97) | 9.88 (4.45)

ADVERSE EVENTS:
Arm/Group | Treatment Modification | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes